CLINICAL TRIAL: NCT06440239
Title: A Phase 1/Phase 2a Study to Evaluate the Safety, Tolerability and Efficacy of PMS-101 Administration in Patients With Burn(s)
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy in Patients With Burn(s)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Primoris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMS-101-A001
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Burns; Burn Degree Second
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): PMS-101
  Interventions: Drug: PMS-101
- Control (Other): Standard of care or treatment
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: PMS-101 — PMS-101
  Arms: Investigational Product
Other: Standard treatment — Standard treatment according to physicians
  Arms: Control

SUMMARY:
For Phase 1, researchers will explore the safety, and tolerability of PMS-101 and determine the recommended Phase 2 dose (RP2D) using the donor site.

For Phase 2a, researchers will compare PMS-101 to a standard-of-care to see if PMS-101 works to treat mid-dermal burns.

DETAILED DESCRIPTION:
Phase 1 is a single arm, open label, non-randomised study designed to assess the safety, tolerability and efficacy of 2 planned dose levels of PMS-101. The decision to continue dosing in Cohort 2(higher level dose) at the planned dosage regimen will be made by the Safety Review Committee (SRC) following the review of the safety and tolerability data of the participants in Cohort 1(lower level dose). The tolerability assessment of all the enrolled participants will be completed to determine the RP2D.

Phase 2a is a double arm, open label, randomised study designed to assess the safety and efficacy of the dose recommended after the tolerability assessments of all participants enrolled in Phase 1 study.

ELIGIBILITY:
Inclusion Criteria:

1. The combined TBSA of all burns is 10% or less.
2. Nonsmoker and must not have used any tobacco products within 2 months prior to Screening.
3. Phase 1 only: Participants with TBSA < 10% who will undergo autologous skin grafting.
4. Phase 2a only: Participants with dermal burns who are within 5 days from the date of wound and will be enrolled.
5. Phase 1 only: Those who have confirmed at least 1 donor wound site with an even distribution of depth and extent of maximum 1% TBSA as judged by the Investigator.
6. Phase 2a only: Those who have confirmed at least 2 dermal burn sites with similar depth and extent of 50 cm2 or more each as judged by the Investigator.

Exclusion Criteria:

1. Those who are allergic to or have experienced hypersensitivity to any components of the IP or its excipients such as gelatin or hyaluronic acid ingredients.
2. Those with the following conditions for burns at the time of Screening in clinical trials:

   1. Those who have suffered chemical or electrical burns (for Phase 2a only).
   2. Persons requiring tracheal intubation or tracheostomy due to severe inhalation burns.
   3. Those with burn wounds accompanied by trauma such as fractures or lacerations.
   4. Persons with purulent infection of burn wounds.
   5. Those who require treatment such as artificial mechanical ventilation, extracorporeal membrane oxygen therapy, or dialysis due to other concomitant diseases or conditions.
3. History of or active bleeding or coagulation diseases (eg, hemophilia, von Willebrand's disease, thrombocytopenia, disseminated intravascular coagulation).
4. History of or active autoimmune diseases (eg, systemic lupus erythematosus, rheumatoid arthritis, Sjögren's syndrome, Behcet's disease, and/or multiple sclerosis.
5. History of or active cardiovascular disease including clinically significant arrhythmias, uncontrolled hypertension, coronary artery disease (CAD), and/or prolonged QT interval (QTc > 450 msec for males and > 470 msec for females).
6. History of or active ischemic, hemorrhagic, or anatomical neurovascular disease including, but not limited to, trans ischemic attack, cerebrovascular accident, arterio-venous malformation, or brain aneurysm.
7. History of or active peripheral vascular disease such as deep vein thrombosis, pulmonary embolism, chronic venous insufficiency, claudication, or lymphedema.
8. History of active pulmonary diseases including chronic obstructive pulmonary disease, pulmonary fibrosis, moderate-to-severe sleep apnea, and moderate-to-severe asthma.
9. Active malignancy, other than local subcutaneous squamous cell and basal cell carcinomas.
10. History of immunosuppressive, chemotherapeutic, or radiation treatment within the last 12 months prior to Screening.
11. History of type 1 diabetes or active type 2 diabetes.
12. History of severe endocrine disorders such as Cushing's disease, hypogonadism, and growth hormone deficiency.
13. History or presence of severe active acute or chronic liver disease (eg, cirrhosis), hepatic insufficiency defined as Child Pugh Class A or higher, nonalcoholic fatty liver disease (NAFLD), nonalcoholic steatohepatitis (NASH), general hepatic disease including serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × the upper limit of normal.
14. Uncontrolled psychiatric disease including major depressive disorder, bipolar, anxiety disorder, or eating disorders such as bulimia.
15. Those with serious diseases or condition that the Investigator believes may affect wound healing, such as a malnourished, clinically significant vitamin and/or mineral deficiencies.
16. Positive test for HIV, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody at the initial Screening Visit.
17. History of systemic active infectious diseases (eg, sepsis, tuberculosis) at the initial Screening Visit.
18. Those who have a history of malignant tumor or lymphoproliferative disease or have received an organ transplant within 5 years of initial Screening Visit.
19. Participants who have received systemic steroids, immunosuppressants, antiplatelet agents or anticoagulants within 1 week before application of this clinical trial drug.
20. History of abnormal wound healing such as keloids or hypertrophic scars.
21. History of significant drug abuse within 12 months prior to Screening or positive urine drug test at Screening.
22. Chronic kidney disease Stages 1 to 5.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Tolerability assessed by dose-limiting toxicity (Phase 1) | Day7, Day9, Day11, Day14, Day17, Day21, Day28, Day56
Time to complete healing of wound site (Phase 2a) | Day7, Day9, Day11, Day14, Day17, Day21, Day28, Day56, Day84

CONTACTS AND LOCATIONS:
Overall Officials: Joanneke Joanneke, Dr, Principal Investigator — The Concord Repatriation General Hospital
Locations (1):
- The Concord Repatriation General Hospital, Sydney, New South Wales, Australia